CLINICAL TRIAL: NCT01933568
Title: Combined Stereotactic Radiotherapy and Conventional Fractionation in Stage II and III Non Small Cell Lung Cancer (NSCLC) With Peripheral Tumors Smaller Than 5 cm
Brief Title: Combined CFRT and SABR in Stage II and III NSCLC With Peripheral Tumors Smaller Than 5 cm.
Acronym: N12HYB
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N12HYB
Record Dates: First submitted 2013-08-28; First posted 2013-09-02 (Estimated); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Inoperable Locally Advanced Non Small Cell Lung Cancer
MeSH Terms: interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiation (Experimental): combined CFRT and SABR with concurrent cisplatin
  Interventions: Radiation: SABR; Drug: Cisplatin

INTERVENTIONS:
Radiation: SABR — combined CFRT and SABR with concurrent cisplatin
Drug: Cisplatin — combined CFRT and SABR with concurrent cisplatin

SUMMARY:
A phase I trial is being conducted in patients with inoperable locally advanced NSCLC to treat with a combination of Conventional Fractionated Radiotherapy (CFRT) on the mediastinal lymph nodes and Stereotactic Ablative Radiotherapy (SABR)on the primary tumor with concurrent chemotherapy. It is hypothesized that this will lead to an increase of local control and overall survival

DETAILED DESCRIPTION:
In locally advanced NSCLC local control has been poor, but with SABR remarkable high local control rates with low toxicity have been reported. Currently stage III and inoperable II NSCLC patients have been treated with IMRT and concurrent chemotherapy at out institute. In this study we will explore the combination of SABR and CFRT with concurrent chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* Cytological or histological proven NSCLC stage III or inoperable stage II, cT1-2a-3N1-3M0 with peripheral tumors < 5 cm (chest wall infiltration is no exclusion criteria if the tumor diameter is < 5 cm).
* Weight loss < 10% in the last three months
* WHO-performance status ≤ 2
* Patients that receive concurrent chemoradiotherapy, with the exception of adriamycin and gemcitabine
* FEV1 and DLCO > 40 % of the age-adjusted normal value
* Minimum required laboratory data bone marrow reserve and hepatic- and renal function
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* Before patient registration, written informed consent must be given according to GCP and national regulations

Exclusion criteria:

* Patients with central tumors < 2 cm of the proximal bronchial tree (Figure 2) or tumors immediately adjacent to mediastinal or pericardial pleura.
* Patients that receive sequential chemoradiotherapy or radiotherapy only.
* Patients with grade 3 dyspnea at baseline (according to CTCAE version 4.03)
* Patients with Pancoast tumors
* Prior radiotherapy treatment to the thorax
* Any contraindications to the administration of thoracic radiotherapy
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-02-28 (Actual); Primary Completion 2018-11-11 (Actual); Study Completion 2018-11-11 (Actual)

PRIMARY OUTCOMES:
The mean-lung dose that is associated with a 15% probability of dose limiting toxicity, defined according to the CTCAE v4; radiation pneumonitis ≥ grade 3 and radiation induced dyspnea ≥ grade 3. | 2 yrs

CONTACTS AND LOCATIONS:
Overall Officials: Heike Peulen, MD, Principal Investigator — The Netherlands Cancer Institute
Locations (1):
- The Netherlands Cancer Institute, Amsterdam, Netherlands

REFERENCES:
- [Derived] Peulen H, Franssen G, Belderbos J, van der Bijl E, Tijhuis A, Rossi M, Sonke JJ, Damen E. SBRT combined with concurrent chemoradiation in stage III NSCLC: Feasibility study of the phase I Hybrid trial. Radiother Oncol. 2020 Jan;142:224-229. doi: 10.1016/j.radonc.2019.07.015. Epub 2019 Aug 17. PMID 31431387